CLINICAL TRIAL: NCT06553430
Title: Effects of an Aerobic Exercise Intervention on Core Symptoms, Executive Functioning, and Quality of Life in Children With Attention Deficit Hyperactivity Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Lingrong Xiao, Principal Investigator, Harbin Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LXiao
Record Dates: First submitted 2024-08-08; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Moderate-intensity aerobic exercise for 30-60 min 3 times per week for 12 weeks and daily physical activity
  Interventions: Behavioral: aerobics exercises
- Control group (No Intervention): daily physical activity

INTERVENTIONS:
Behavioral: aerobics exercises — Moderate-intensity aerobic exercise for 30-60 min 3 times per week for 12 weeks
  Arms: Intervention group

SUMMARY:
Selecting a maternal and child healthcare hospital in Shenzhen City, Guangdong Province, 50 cases of ADHD children as the study subjects, according to the inclusion and exclusion criteria to screen the eligible study subjects, introduction of the purpose and process of the study, informed consent to enrolment, the children were divided into the intervention group and the control group. The experimental group used aerobic exercise, while the control group was given daily physical activity, and general information questionnaires, Conners Parental Symptom Questionnaire, SNAP-IV scale, Stroop Colour Word Test, Rey Complex Graphics Test, Connection Test, Children's Depressive Disorder Self-assessment Scale, Children's Anxious Mood Disorder Screening Scale, Children's Quality of Life Universal Core Scale, and Children's Executive Functioning Questionnaire were assessed.

DETAILED DESCRIPTION:
Purposive sampling method was used to select a maternal and child healthcare hospital in Shenzhen City, Guangdong Province, 50 cases of ADHD children as the study subjects, according to the inclusion and exclusion criteria to screen the eligible study subjects, introduction of the purpose and process of the study, informed consent to enrolment, the children were divided into age, gender, clinical typing, medication use, family proximity, Conners scores and SNAP-IV scores matching the intervention group and the control group. The experimental group used aerobic exercise, while the control group was given daily physical activity, and general information questionnaires, Conners Parental Symptom Questionnaire, SNAP-IV scale, Stroop Colour Word Test, Rey Complex Graphics Test, Connection Test, Children's Depressive Disorder Self-assessment Scale, Children's Anxious Mood Disorder Screening Scale, Children's Quality of Life Universal Core Scale, and Children's Executive Functioning Questionnaire were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Children clinically diagnosed with ADHD;
* 7-14 years old;
* Combined Raven's Test ≥ 80;
* Not participating in any treatment other than drug therapy;
* The body can participate in sports training;
* The type of family intimacy is intimate or above;
* Voluntarily participate and sign an informed consent form

Exclusion Criteria:

* Children with a history of epileptic seizures;
* Children with other mental or motor disorders;
* Children with visual impairments;
* Using other psychotropic drugs;
* Have other comorbidities;
* Merge other serious chronic diseases (such as severe heart, brain, kidney, lung, etc.), tumors, etc

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
ADHD core symptoms | Immediately after the intervention
  The Conners Parental Symptom Questionnaire for core symptoms. There are a total of 48 items, including six factors. They are scored on a scale of 0-3, with 0 indicating no problem; 1, occasionally or slightly; 2, frequent or severe; 3, always or very serious. The factor score is the average score of the items within the factor, and the higher the score, the more severe the symptom. The SNAP-IV for ADHD children's inattention and hyperactivity/impulsivity. This scale consists of 26 items and consists of three subscales. Each item is rated on a four point scale from 0 to 3: 0, "never or rarely"; 1, "sometimes"; 2, "often"; 3, 'very common'. The average score of each subscale is the ratio of the total score of the obtained items to the number of items included. Scores from 0-1 are considered normal, 1.1-1.5 are critical, 1.6-2 are moderate, and>2 are severe. The higher the total score and subscale score, the more severe the damage to the core symptoms of ADHD.

SECONDARY OUTCOMES:
executive function | Immediately after the intervention
  Stroop color-word test for Inhibitory control, Rey-Osterrieth Complex Figure for working memory, Trail Making Test for cognitive flexibility and Questionnaire of Executive Functioning Scale for total executive function. The Questionnaire of Executive Functioning Scale consists of 36 items and 8 factors including attention concentration, working memory, self-regulation, theory of mind, flexible switching, impulse suppression, plan initiation, and emotion regulation. All items are rated on a 4-point scale from 1 (never) to 4 (always). The higher the score, the worse the performance of the execution function.
quality of life | Immediately after the intervention
  The Pediatric Quality of Life Inventory Version 4.0 Generic CoreScales to measure ADHD children's quality of life. The scale has 23 items, including four dimensions: physiological function, emotional function, social function, and role function. Each item is scored on a Likert 5-point scale, and the total score of the scale is equal to the sum of the scores of each item. The higher the score, the better the quality of life.
mental health | Immediately after the intervention
  Depression Self-Rating Scale for Children to measure depression. There are a total of 18 items, rated on a 0-2 scale, with 0 indicating no symptoms, 1 indicating occasional symptoms, and 2 indicating frequent symptoms. The sum of each item is the total score, with higher scores indicating more severe depression, and a total score greater than 14 indicating possible depression. Screen for Child Anxiety Related Emotional Disorders to measure anxiety. There are a total of 41 items consisting of 5 factors, namely somatic symptoms/panic, generalized anxiety, dissociative anxiety, social phobia, and school phobia. Each item is rated on a scale of 0-2, where 0 indicates no such symptoms, 1 indicates partial presence, and 2 indicates frequent presence. The higher the score, the more severe the anxiety level. A total score of more than 23 on the scale may indicate a significant state of anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Nanshan Maternal and Child Health Hospital, Guangzhou, Shenzhen, China